CLINICAL TRIAL: NCT05019599
Title: Exploring the Role of Low Protein Diet on the Gut Microbiome, Related Metabolites and Renal Function in Chronic Kidney Disease
Brief Title: Low Protein Diet, Gut Microbiome and Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IWW-0008
Record Dates: First submitted 2021-01-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Intervention Model Description: nutritional intervention with low protein diet (< 0.8 G protein/kg body weight/day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal controls (No Intervention): subjects with normal renal function
- CKD_Low protein diet (Experimental): CKD patient with low protein diet (<0.8g/kg/BW)
  Interventions: Other: low protein diet
- CKD_normal protein diet (Active Comparator): CKD patient with normal protein diet
  Interventions: Other: low protein diet

INTERVENTIONS:
Other: low protein diet — Low protein diet (<0.8g/kg/BW/day)
  Arms: CKD_Low protein diet; CKD_normal protein diet

SUMMARY:
Chronic kidney disease (CKD) is a worldwide public health dilemma because of close association with multiple comorbidities, demanding high cardiovascular events, mortality and expensive medical cost. Novel and effective therapeutic measures remain urgently needed to reduce burden and impact of disease. Advanced renal failure can profoundly alter the biochemical milieu of the gastrointestinal tract leading to a leak gut. Application of 16s rRNA gene analysis identified an increase of Clostridia, Actinobacteria, and Gammaproteobacteria in hemodialysis patients and decrease of Bifidobacterium and lactobacillus in peritoneal patients. This altered microbiome consequently affect production of indole or phenol derived uremic toxins leading to renal damage. Our preliminary results indicated reduced number and diversity of intestinal microbes CKD patients compared to normal. Different dietary nutrients can affect the gut microbiome and derive several deleterious metabolites leading to metabolic disarrangement. Clinically, low-protein diet should be prescribe to renal patients to preserve renal function and high fat content are usually recommended to avoid caloric malnutrition to dietary restriction. The changes of diet-microbiome-metabolite interaction are large unknown with this dietary manipulation. The aims of this study is to determine the renal progression-associated gene and taxonomic alterations bymetagenome-wide association studies and the functional characterization of gut microbiome in CKD patients receiving different low-protein or high-fat diets. The results of the study will provide insight on the exact role of dietary manipulation in CKD patients from gut-renal cross talk.

ELIGIBILITY:
Inclusion Criteria:

1. . Patients aged 30-90 years with diagnosis of CKD (defined as abovementioned).
2. . Sign the inform consent and agree to participate in this study.
3. . Compliant to low protein diet (defined as protein intake <0.8 g/Kg/day) for 4 weeks assessed by 24h urine urea estimates, before enrollment

Exclusion Criteria:

1. . History of any malignancy, liver cirrhosis, intestinal operation, irritable bowel syndrome, cardiovascular disease (defined as myocardial infarction, documented Q wave on EKG, unstable angina, coronary artery disease with stenosis > 75%, congestive heart failure with Ejection Fraction < 50% and cerebrovascular disease) in the past 3 months.
2. . History of or infection disease requiring admission in the past 3 months or, concomitant antibiotics use.
3. . Concomitant use of probiotics or prebiotics.
4. . Pregnancy.
5. . Renal transplant recipients.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
change of gut microbiota | 3 months
  change of relative abundance of microbes
change of host metabolite concentration | 3 months
  change of concentration of serum metabolomic profile
change of renal function | 3 months
  serum creatinine, estimated glomerular filtration rate or urine total protein

CONTACTS AND LOCATIONS:
Overall Officials: I Wen Wu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu IW, Lee CC, Hsu HJ, Sun CY, Chen YC, Yang KJ, Yang CW, Chung WH, Lai HC, Chang LC, Su SC. Compositional and Functional Adaptations of Intestinal Microbiota and Related Metabolites in CKD Patients Receiving Dietary Protein Restriction. Nutrients. 2020 Sep 12;12(9):2799. doi: 10.3390/nu12092799. PMID 32932711
- See also: Related Info — https://res.mdpi.com/d_attachment/nutrients/nutrients-11-03006/article_deploy/nutrients-11-03006.pdf